CLINICAL TRIAL: NCT06244173
Title: Clinical and Laboratory Parameters of Myelodysplastic Syndromes at Upper Egypt
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed Abdel-baset, lecturer of internal medecine, Sohag University
Other Study IDs: Soh-Med-23-09-8PD
Record Dates: First submitted 2023-10-04; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to assess clinical & laboratory parameters of adult Egyptian myelodysplastic syndrome patients in upper Egypt, its correlation with disease-free survival, overall survival (OS) and acute leukemia transformation.

DETAILED DESCRIPTION:
The aim of this study is to assess clinical & laboratory parameters of adult Egyptian myelodysplastic syndrome patients in upper Egypt, its correlation with disease-free survival, overall survival (OS) and acute leukemia transformation.

Materials and methods:

This study will be conducted in Sohag University Hospital and Assuit University Hospitals on available number of newly diagnosed patients with MDS according to the diagnostic criteria proposed by the WHO in 2016 .

full history taking, clinical assessment and certain laboratory investigations are conducted to every patient enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* De novo MDS according to WHO criteria diagnosis 2016

Exclusion Criteria:

* MDS on top of AML

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: cases of Denovo MDS attending to Sohag Univeristy hospital and Assuit University hospitals
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
overall survival | baseline
  analysis of collected data

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa abdelbaset, MD, Principal Investigator — faculty of medicine - Sohag university
Locations (1):
- Sohag univeristy hospitals, Sohag, Egypt